CLINICAL TRIAL: NCT06737705
Title: Efficacy and Safety Study of Baricitinib for Respiratory Injury in Patients With Intracerebral Hemorrhage
Brief Title: Baricitinib for Respiratory Injury in Patients With Intracerebral Hemorrhage
Acronym: BRIGHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: De-zhi Kang (Other)
Collaborators: Fujian Medical University (Other); Tianjin Medical University General Hospital (Other)
Responsible Party: Sponsor-Investigator, De-zhi Kang, Prof., First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRCTA, ECFAH of FMU [2024] 556
Record Dates: First submitted 2024-12-10; First posted 2024-12-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Intracerebral Hemorrhage; Acute Lung Injury(ALI)
Keywords: Intracerebral Hemorrhage; Acute Lung Injury; Baricitinib
MeSH Terms: conditions — Cerebral Hemorrhage; Acute Lung Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard care (No Intervention): Standardized treatment for respiratory protection and/or ALI after ICH according to the related guidelines.
- Standard care plus Baricitinib (Experimental): Besides standardized treatment (background therapy) for respiratory protection and/or ALI after ICH according to the related guidelines, participants will receive additional baritinib administration.
  Interventions: Drug: Baritinib

INTERVENTIONS:
Drug: Baritinib — Participants will receive additional baritinib administration with 4-mg dosage once daily (QD) for consecutive 14 days after randomization (adjusted dosage of 2-mg QD for participants with eGFR between 30-60 mL/min/1.73m^2).
  Arms: Standard care plus Baricitinib

SUMMARY:
This study is an investigator-initiated, prospective, randomized, open-label, blind end-point (PROBE) phase-2 clinical trial, to preliminarily evaluate the efficacy and safety of baritinib for the treatment of acute lung injury (ALI) after spontaneous intracerebral hemorrhage (ICH). Approximately 100 patients from different geographic sites across China will be recruited and randomized to 2 parallel arms in a 1:1 ratio to the intervention arm or control arm. The study will compare early additional baritinib 4-mg once daily (QD) administration to control arm with standardized treatments (background therapy), as novel agents for ALI in aimed subjects in immunological approach; and provide cortical evidence for further phase-3 clinical trials. The trial will be across up to approximately 15-month scope (12-month enrollment period and 3-month follow-up period). One independent Data and Safety Monitoring Board (DSMB) will actively monitor interim data in all stages to make recommendations about early study closure or changes to study protocol.

ELIGIBILITY:
* Inclusion criteria

  1. Participant (or legally authorized representative) who gives informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol;
  2. Are male or female patients from 18 years of age (inclusive), at the time of enrollment;
  3. Have acute, spontaneous, primary, supratentorial intracerebral hemorrhage (ICH), confirmed by head CT scan, at the time of enrollment;
  4. Complicated with acute lung injury (ALI), confirmed by chest CT scan, at the time of enrollment.
* Exclusion criteria

  1. Have cerebellar or brainstem ICH;
  2. Have secondary ICH due to known or suspected structural abnormality in the brain, i.e., trauma, aneurysm, arteriovenous malformation, tumor;
  3. Have severe cerebral comorbidities, i.e., historical severe stroke, hydrocephalus, epilepsy;
  4. Have known advanced dementia or significant pre-stroke disability (modified Rankin Scale score of > 1);
  5. Have comorbidities might result in ALI, i.e., interstitial lung disease, chronic obstructive pulmonary disease, lung tumor, asthma, chronic respiratory failure, chronic heart failure;
  6. Have severe immunosuppression, defined as neutropenia (absolute neutrophil count < 1.0×10^9 cells/L) or lymphopenia (absolute lymphocyte count < 0.2×10^9 cells/L);
  7. Have chronic autoimmune disease, i.e., neuromyelitis optica spectrum disorders, multiple sclerosis, rheumatoid arthritis, systemic lupus erythematosus;
  8. Have ever received attenuated live vaccination or immunological treatments (see below) within 4 weeks prior to the enrollment, or intend to receive measures above;

     * Cytotoxic treatments: cyclophosphamide, methotrexate, sulfasalazine, leflunomide, etc.;
     * Biological treatments: adalimumab, infliximab, etanercept (TNF-α inhibitors), tocilizumab (anti-IL-6), secukinumab (anti-IL-17), etc.;
     * Baricitinib and other JAK inhibitors: tofacitinib, abrocitinib, etc.;
     * Other treatments: convalescent plasma or intravenous immunoglobulin (IVIg), corticosteroids with dosage over alternative purpose, etc.;
     * Note: Non-steroid anti-inflammatory drugs (NSAID) are allowed;
  9. Have current or historical infections within 2 weeks prior to the enrollment, i.e., pneumonia, SARS-CoV-2 infections, current active tuberculosis; or have ever received antibiotics within 2 weeks prior to the enrollment;
  10. Have contraindications for baricitinib, i.e., severe anemia (hemoglobulin < 80g/L), decompensated kidney disease (eGFR < 30mL/min/1.73m^2), or severe liver injury with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times ULN;
  11. Have a current diagnosis of active malignancy, history of deep vein thrombosis (DVT) and/or pulmonary embolism (PE) within 12 weeks prior to the enrollment or have a history of recurrent DVT/PE (≥ 2 times in total), which could constitute a risk when taking baricitinib in the opinion of the investigator;
  12. Are unlikely to finish the whole course of baricitinib administration in the opinion of the investigator (anticipated death or discharge);
  13. Are pregnant, or intend to become pregnant or breastfeed during the study;
  14. Are recruited for any other clinical trials;
  15. Are unsuitable for inclusion in the study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
The score shift on the radiologic scoring system for lung injury involvement from baseline to day 14 after randomization | From baseline to day 14 after randomization
  This radiologic scoring system for lung injury involvement was assessed with the chest CT scan, ranging from 0 to 10. The lower score indicated less lung injury while the higher represented more.

SECONDARY OUTCOMES:
The modified Rankin Scale (mRS) score at day 90 after randomization | At day 90 after randomization
  The mRS ranged from 0 to 6 and usually was adopted for neurological assessment. The lower score indicated favorable outcome while the higher represented worse or even death.
Time from randomization to the day of at least 1-point improvement on the National Institute of Allergy and Infectious Disease Ordinal Scale (NIAID-OS) | From randomization to the presence of clinical end-point (NIAID-OS improvement ≥ 1 point, discharge, or death) or the end of observation (up to 90 days after randomization), whichever comes first
  The NIAID-OS was for respiratory assessment, ranging from 1 to 8 in the original version. In this trial, the NIAID-OS was measured ranging from 3 to 8 (inclusive). The lower score indicated mild symptoms while the higher represented more critical or even death.
Peripheral blood interleukin-6 (IL-6) level at day 14 after randomization | At day 14 after randomization
Peripheral blood interleukin-8 (IL-8) level at day 14 after randomization | At day 14 after randomization
Peripheral blood C-reactive protein (CRP) level at day 14 after randomization | At day 14 after randomization

CONTACTS AND LOCATIONS:
Overall Officials: De-zhi Kang, M.D., Principal Investigator — First Affiliated Hospital of Fujian Medical University; Ying Fu, Ph.D., Study Director — First Affiliated Hospital of Fujian Medical University
Locations (6):
- China (6):
  - The Southwest Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - Liaocheng People's Hospital, Liaocheng Brain Hospital, Liaocheng, Shandong
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided